CLINICAL TRIAL: NCT01673113
Title: Characterization of Transient Alterations of Cutaneous Sensory Nerve Function by Cryolipolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Professor, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-P-001380
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Adiposity
Keywords: cryolipolysis, sensory nerve function, Zeltiq
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryolipolysis (Experimental): All subjects were randomized to have either the left of right flank treated with single the Zeltiq CoolSculpting Device, which is an FDA approved cooling device used for non-invasive and selective reduction of fat around the flanks. Sensory testing was done before and after the procedure.
  Interventions: Device: Zeltiq CoolSculpting device
- Control (No Intervention): All subjects were randomized to have either the left of right flank treated with single the Zeltiq CoolSculpting Device. The untreated flank served as the internal control for each subject.

INTERVENTIONS:
Device: Zeltiq CoolSculpting device — This is an FDA approved cooling device used for non-invasive and selective reduction of fat around the flanks, an area commonly referred to as the "love handles."
  Arms: Cryolipolysis

SUMMARY:
Cryolipolysis with Zeltiq CoolSculpting device is a novel method of non-invasive fat removal. The technique works by application of cold plates to the skin surface for a single cooling cycle lasting 60 minutes, after which a cold-induced inflammatory panniculitis leads to selective loss of fat. There is no histologic evidence of necrotic or inflammatory damage to skin or nerves, however a single small human study has reported prolonged temporary altered sensation (hypoesthesia) in the area of cryolipolysis procedure. This hypoesthesia seen in about 2/3 of patients, is completely reversible, lasts up to 8 weeks after treatment, and suggests that cooling under these conditions can temporarily alter sensory nerve function.

The purpose of this study is to further characterize the reversible cutaneous sensory function alteration after cryolipolysis with Zeltiq CoolSculpting device. Using multiple modalities of sensory nerve function we hope to elucidate the details of cryolipolysis induced sensory nerve alteration.

DETAILED DESCRIPTION:
Study design We undertook an open-label, prospective study at the Massachusetts General Hospital (MGH) (Boston, USA) between December 2012 and July 2013. The study was approved by the MGH Institutional Research Board and was registered at ClinicalTrials.gov (NCT01673113). Written, informed consent was obtained from all participants prior to participation in the study. The study conformed to the standards set by the Declaration of Helsinki and Good Clinical Practice Guidelines.

Eleven healthy subjects were enrolled in the study. They were randomized to have either the left or right flank treated with a single cycle of cryolipolysis. Baseline measurement of sensory function was evaluated using QST at the treated and control (untreated) flank for each subject. Histamine iontophoresis was used to evaluate itch duration and intensity on the treated and control flank for each subject. All sensory function testing, including responses to histamine-induced itch, were assessed at 48-72 hours, and Day 7, 14, 21, 35 and 56 post-treatment. In 6 subjects, skin biopsies (3 mm diameter) for histological analysis of nerve fiber density at the treated flank were taken at baseline, 48-72 hours, Day 21 and 56 post-treatment.

Cryolipolysis procedure All subjects received cryolipolysis treatment to the flank above the iliac crest, on one side of the body. The untreated (contralateral) flank served as the control throughout the study. Subjects were randomized to have right or left flank treated and randomization was achieved with a computer-generated randomization code. The treatment site was identified, assessed and marked by a single, unblinded investigator. The sensory testing site within the flanks was marked and registered using a transparent plastic sheet, aligned using cutaneous landmarks including nevi or scars, and photographed with the subject in a standard position, to ensure that the same area was tested on follow-up visits.

Cryolipolysis was performed using an EzApp6.3 applicator (CoolScultping, Zeltiq Aesthetics Inc, Pleasanton USA) and standard settings at cooling intensity factor (CIF) of 41.6, corresponding to heat transfer of -73mW/cm2, applied for one hour.

Quantitative sensory testing (QST) The QST protocol consisted of a series of 7 sensory tests. The QST procedure started with the evaluation of mechanical followed by thermal thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18-65 years old, male or female with visible adiposity on the flanks (love handles) and no weight changes exceeding 10lb during the preceding month.
* Willingness to participate in the study
* Informed consent agreement signed by the subject
* Willingness to follow the treatment schedule and post treatment care requirements
* Willingness to have skin biopsy done
* No history of allergy to lidocaine or any other anesthetics.

Exclusion Criteria:

* Subject has a history of nerve problems, neuropathy
* Subject who has recently undergone liposuction or another weight loss procedure, had a history of subcutaneous injections into the area of intended treatment within the preceding 6 months.
* Subjects with history of diabetes
* Subjects with a BMI of 30 or greater
* Subject has an infection, surgical scars or other dermatologic condition in the area to be treated
* Subject has known cold sensitivity disorders including Raynaud's phenomena, cold urticaria, cryoglobulinemia, or cold induced hemoglobinuria
* Women who are pregnant or intending to become pregnant in the following 9 months; women who are lactating or had been lactating in the prior 9 months.
* Subject is immunosuppressed
* Subject is unable to comply with treatment, home care or follow-up visits
* Subject has a history of vitiligo
* Subject has a history of keloid formation
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.
* Subject taking anticoagulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Rox Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garibyan L, Cornelissen L, Sipprell W, Pruessner J, Elmariah S, Luo T, Lerner EA, Jung Y, Evans C, Zurakowski D, Berde CB, Rox Anderson R. Transient Alterations of Cutaneous Sensory Nerve Function by Noninvasive Cryolipolysis. J Invest Dermatol. 2015 Nov;135(11):2623-2631. doi: 10.1038/jid.2015.233. Epub 2015 Jun 22. PMID 26099028
- See also: the published paper — http://www.ncbi.nlm.nih.gov/pubmed/26099028

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 subjects were randomized to have either left or right flank treated. The untreated flank served as the internal control for each subject.
Units Other Than Participants: flanks
Groups:
- Treatment: Subjects were randomized to have either left or right flank treated with cryolipolysis.
- Control: The untreated flank of each subject served as internal control.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 11; 11 flanks | 11; 11 flanks
Completed | 11; 11 flanks | 11; 11 flanks
Not Completed | 0; 0 flanks | 0; 0 flanks

BASELINE CHARACTERISTICS:
Population: BMI of <30 kg/m^2
Units Other Than Participants: flanks
Groups:
- Treatment: Subjects were randomized to have right or left flank treated with Zeltiq CoolSculpting device
- Control: The untreated flank of each subject served as the internal control.
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (flanks) | 11 | 11 | 22
Age, Categorical [Count of Units; unit: flanks]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: flanks]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: flanks]
  United States | 11 | 11 | 22
BMI of <30 [Count of Units; unit: flanks] | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Vibration Detection Threshold (VDT)
Description: VDT was evaluated using a computerized vibrometer with 1cm2 contact probe placed perpendicularly on the skin (TSA-II, Medoc Inc., Ramat Yishai, Israel). This device gradually increased the vibration magnitude until the subject pressed a "stop" button to indicate when they first felt the vibration. This test was repeated 8 times. The values presented in the data table were averaged over all repeats.
Time Frame: within 48-72 hours after treatment
Population: 11 subjects were randomized to have right or left flank treated with cryolipolysis. The untreated flank served as the internal control.
Measure: Mean (95% Confidence Interval); unit: (um/sec)
Units Other Than Participants: flanks
Groups:
- Treatment: Cryolipolysis treated flanks had vibration sensory testing done within 48-72 hours after treatment.
- Control: Untreated flanks of each subject had vibration sensory testing done within 48-72 hours after treatment.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 11 | 11
Number analyzed (flanks) | 11 | 11
(um/sec) | 26.3 [20.9 to 31.7] | 19 [13.6 to 24.4]

2. Secondary Outcome: Mechanical Detection Threshold (MDT)
Description: MDT was evaluated using von Frey Filaments. The up-down method, which evaluates the threshold force for appearance and disappearance of a touch sensation reported by the subject, was used until 3 values were obtained. The values presented in the data table were averaged over all repeats.
Time Frame: 48-72 hours post treatment
Population: 11 subjects were randomized to have right or left flank treated with cryolipolysis and the untreated flank served as internal control.
Measure: Median (Inter-Quartile Range); unit: grams
Units Other Than Participants: flanks
Arm/Group | Treatment | Control
Number analyzed (Participants) | 11 | 11
Number analyzed (flanks) | 11 | 11
grams | 0.87 [0.4 to 1.27] | 0.4 [0.21 to 0.93]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the duration of the study.
Arm/Group | Cryolipolysis
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes